CLINICAL TRIAL: NCT05566769
Title: Performance and Safety of a Digital Tool for Unsupervised Self-assessment of Neuromyelitis Optica Spectrum Disorder
Brief Title: Performance and Safety of a Digital Tool for Unsupervised Self-assessment of NMOSD
Acronym: OPTIS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ad scientiam (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: OPTIS
Record Dates: First submitted 2022-09-07; First posted 2022-10-04 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Neuromyelitis Optica
Keywords: NMO; NMOSD; Neuromyelitis optica; Neuromyelitis optica spectrum disorder
MeSH Terms: conditions — Neuromyelitis Optica

STUDY DESIGN:
Intervention Model Description: One group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- NMOSDCopilot (Experimental): Performance of digital tests and standard test in clinic at D0 and M6 Use of NMOSDCopilot at-home in between visits during 12 months
  Interventions: Device: NMOSDCopilot smartphone application

INTERVENTIONS:
Device: NMOSDCopilot smartphone application — NMOSDCopilot includes active tests for walking, cognition, dexterity and vision, and e-questionnaires related to pain, fatigue, quality of life, bladder and bowel dysfunction, depression

SUMMARY:
NMOSDCopilot is a digital tool developed for the self-assessment of Neuromyelitis Optica Spectrum Disorder symptoms that impact patients' functioning and quality of life. It has been co-designed with the help of patient advocacy groups, NMOSD patients and medical experts. It includes a smartphone-based application for patients, connected to a web portal developed for healthcare professionals (HCSPs). The patient application is composed of vision, walking, cognition, and dexterity e-active tests inspired by clinical standards, as well as e-questionnaires. The HCP web portal is a desktop-based software that allows HCPs to access the results generated via the patient application and facilitates remote monitoring of patients' symptoms.

The objectives of this study are to validate the accuracy, reliability and reproducibility of the unsupervised at-home self-assessment of symptoms on the patient's smartphone versus the standard in-clinic testing, as well as to evaluate the safety of use of the tool, its usability, and satisfaction towards the patient application among NMOSD patients, and the HCP web dashboard among HCPs.

ELIGIBILITY:
Inclusion Criteria:

* Aged over 18 years old
* NMOSD as defined by the 2015 international consensus diagnostic criteria (AQP4+ only)
* With NMOSD treatment (treatment must be unchanged since 6 months before enrollment, and 1 month for analgesics, antidepressants, neuroleptics)
* EDSS =< 7
* With no evidence of relapse in the past 3 months before enrollment
* Who have read the information sheet and signed the informed consent form
* Able to use a smartphone
* Owns a personal smartphone which version is above 13 for IOS and 8 for Android included
* Able to read language in which the mobile application is available and able to understand pictograms

Exclusion Criteria:

* Evidence of neurologic, rheumatologic or psychiatric disorder other than NMOSD, including but not limited to major head trauma, seizures or systemic medical diseases that are likely to affect cognitive, upper limb or lower limb functioning
* Pregnant and nursing women
* Person under guardianship or curatorship
* Bedridden patients or patients with a daily activity of less than 2 hours per day
* Current drugs or/and alcohol abuse that could influence performance on the tests (clinician's judgment)
* Subject has participated in another clinical study within the previous 30 days of screening or is currently participating in another study that, in the opinion of the Investigator, might interfere with the participant's full participation in the study or confound the assessment of the participant or outcome of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Estimated)
Dates: Start 2023-11-03 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
To compare results obtained with unsupervised at-home e-active tests and the corresponding supervised in-clinic standard tests, test to test | Standard tests results at Baseline versus e-active tests results at D0 + 7 days
  Pearson correlation coefficient (or Spearman's rank-order correlation depending on the data distribution) between e-active tests at day 7 versus standard tests at baseline

SECONDARY OUTCOMES:
To assess reproducibility between in-clinic and at-home e-active tests | Baseline, day 7, month 6 - 7 days, month 6
  Pearson correlation coefficient (or Spearman's rank-order correlation depending on the data distribution) between e-active tests at day 7 versus standard tests at baseline and between and month 6 and month 6- 7days
To assess test-retest reliability of at-home e-active tests | Month 1, month 2, month 3, month 4, month 5
  Intraclass correlation coefficient of e-active tests
To compare results obtained with in-clinic e-active tests and in-clinic standard tests, test to test | Baseline, month 6, month 12
  Pearson's correlation coefficient of inc-clinic e-active tests and in-clinic standard tests
To assess the adverse events related to of the mobile application use. | through study completion, 21 months
  descriptive analysis of adverse events (AEs) related to the use of the application.
To assess pain | Month 3, month 6, month 12
  Pain Visual Analogue Scale (0-100) higher score meaning a worse outcome
To assess fatigue | Month 3, month 6, month 12
  Modified Fatigue Impact Scale 5 (0-20) higher score meaning a worse outcome
To assess bladder control | Month 3, month 6, month 12
  Bladder Control Scale (0-22) higher score meaning a worse outcome
To assess bowel control | Month 3, month 6, month 12
  Bowel Control Scale (0-22) higher score meaning a worse outcome
To assess depression | Month 3, month 6, month 12
  Patient Health Questionnaire-8 (0-12) higher score meaning a worse outcome
To assess quality of life | Baseline, month 6, month 12
  p-value of multivariate analysis for non-parametric data
To assess disability | Baseline, month 6, month 12
  Expanded Disability Status Scale (0-10), higher score meaning a worse outcome
To assess satisfaction and user experience with the smartphone application and the web dashboard | Through study completion, 21 months
  Descriptive analysis of satisfaction and user experience questionnaires (System Usability Scale (1-100) higher score meaning a better outcome)
To assess at-home compliance and adherence to the patient application | Through study completion, 21 months
  Descriptive analysis of the mobile application's adherence data (number of completed questionnaires, number of sessions performed etc.).
To compare results obtained with at home MVT and in-clinic OCT-scan | Through study completion, 21 months
  The Pearson's correlation coefficient will be used to assess the relation between MVT e-active test at D0 +7 (home) versus standard OCT-scan test at D0 (in clinic). The minimum coefficient to reach is 0.65 to show that low contrast visual acuity measurement is associated with. RNF & GCIP layer thickness

CONTACTS AND LOCATIONS:
Locations (22):
- United States (10):
  - University of Southern California, Los Angeles, California
  - University of California Davis Health, Sacramento, California
  - University of south Florida, Tampa, Florida
  - NorthShore University HealthSystem, Evanston, Illinois
  - Johns Hopkins Outpatient Center (now called Levi Watkins, Jr., M.D., Outpatient Center), Baltimore, Maryland
  - Massachussets General Hospital, Boston, Massachusetts
  - Washington University in St. Louis, Washington, Missouri
  - CC Lou Ruvo Center for Brain Health, Las Vegas, Nevada
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Oklahoma Medical Research Foundation, Oklahoma City, Oklahoma
- France (8):
  - Hôpital Roger Salengro, Lille
  - CHU Marseille - La Timone, Marseille
  - CHU de Montpellier, Montpellier
  - Hopital Pasteur 2, Nice
  - Hopital La Pitié Salpétrière, Paris
  - CHU Rouen, Rouen
  - Hopital de Hautepierre, Strasbourg
  - CHU Toulouse - Hôpital Purpan, Toulouse
- Germany (4):
  - Universitätsklinikum Carl Gustav Carus, Dresden
  - Universitätsklinik Essen, Essen
  - University Munich, Munich
  - Hopital Rechts der Isar der Technischen Universitat Munchen, Munich

IPD SHARING:
Plan to Share IPD: No